CLINICAL TRIAL: NCT04845828
Title: Prospective Randomized Comparison of Sentinel Lymph Node Mapping Using Indocyanine Green and Conventional Pelvic Lymph Node Dissection in Clinical Stage I-II Endometrial Cancer
Brief Title: Randomized Comparison Between Sentinel Lymph Node Biopsy and Lymph Node Dissection in Early Stage Endometrial Cancer
Acronym: SELYE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, MD, PhD, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KGOG 2029
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Endometrial Cancer
Keywords: Sentinel lymph node mapping; Indocyanine green; Fluorescent camera; Lymph node dissection; Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sentinel lymph node mapping (Experimental): The group composed of patients who undergo sentinel lymph node mapping
  Interventions: Procedure: Sentinel lymph node mapping
- Routine lymph node dissection (Active Comparator): The group composed of patients who undergo routine pelvic lymph node dissection
  Interventions: Procedure: Routine lymph node dissection

INTERVENTIONS:
Procedure: Sentinel lymph node mapping — Laparoscopic or robotic hysterectomy with/without bilateral salpingo-oophorectomy 2. Inject 1.25 mg/ml of ICG and a total of 6ml into the cornual area (0.5-1 cm deep) of the uterus. And then inject 1 ml of mucous membrane (1-3 mm deep) and 1 ml of substrate (1-2 cm deep) into the cervix, and a total of 4 ml in each direction of 3 and 9 o'clock.
  3. Sentinel lymph node is excised
  Other Names: Indocyanine green; Fluorescent camera
  Arms: Sentinel lymph node mapping
Procedure: Routine lymph node dissection — 1. Laparoscopic or robotic hysterectomy with/without bilateral salpingo-oophorectomy
  2. Lymph node detection is performed.
  Arms: Routine lymph node dissection

SUMMARY:
Through this clinical trial, the investigators aim to verify the usefulness and stability of sentinel lymph node mapping in endometrial cancer of clinical stage I-II.

DETAILED DESCRIPTION:
The standard treatment for endometrial cancer is total hysterectomy and bilateral salpingo-oophorectomy, peritoneal cytology, and lymph node dissection. Pelvic lymph node dissection helps to set accurate staging and adjuvant therapy group, but it has never been proven to have therapeutic effects by itself. According to the results of two recent randomized clinical trials, routine pelvic lymph node dissection in early stage endometrial cancer doesn't improve survival rates.

Routine pelvic lymph node detection can cause complications in a large number of patients and is associated with poor quality of life. Therefore, it is important to develop a method that can check the status of the lymph node in a less invasive way. Efforts have been made to preserve other lymph nodes with significantly less potential for metastasis through less invasive methods, reducing lymph edema and complications such as bleeding and nerve damage caused by excessive surgery.

Sentinel lymph node dissection is used as a standard treatment for breast cancer and malignant melanoma, and efforts to develop it have recently continued in endometrial cancer and cervical cancer. A SENTICOL study conducted in cervical cancer patients showed a false-negative rate of 0% when both were monitored lymph node dissection. In addition, unlike routine pelvic lymph node dissection, ultra-staging through 0,2mm gas intercepts allow additional detection of less than 2mm of microtransfer or less than 0.2mm of independent tumor cells that have not been found before. In a recent large-scale prospective study of endometrial cancer, sentinel lymph node mapping using indocyanine green and fluorescent imaging was successful at 86%, and sensitivity (patient-by-patient analysis) reported 100% in diagnosis of lymph node metastasis.

As laparoscopic and robotic surgery account for most of the treatment of endometrial cancer patients, a good environment is created for monitoring lymph node exploration using ICG, and sensitivity and detection rate seem to have improved compared to the previous method. However, there has been no prospective study on the effects of patient clinical prognosis, such as a standard treatment, pelvic lymph node resection, and disease-free survival rate, and overall survival rate, so a prospective study is essential. The investigators compare survival rates in the group that does sentinel lymph node mapping and routine pelvic lymph node detection in endometrial cancer in clinical stage I-II.

ELIGIBILITY:
Inclusion Criteria:

1. 20 ~ 80 years old female
2. histologically diagnosed endometrial cancer that has never been treated before.
3. histological type :endometrioid, mucinous, serous, clear cell, uindifferentiated, dedifferentiated, mesonephric adenocarcinoma, mesonephric-like adenocarcinoma, carcinosarcoma, and mixed type
4. histological grade : FIGO grade 1, 2, 3
5. Presumed FIGO stage I-II
6. Planed for laparoscopic or robotic hystererctomy and lymph adenectomy
7. Largest pelvic or para-aortic lymph node diameter = or < 15 mm in short axis on MRI
8. ECOG performance status 0-2
9. ASA PS 0-2
10. WBC ≥ 3,000/mm3, Platelets ≥ 100,000/mm3, Creatinine ≤ 2.0 mg/dL ,Bilirubin ≤ 1.5 x institutional upper limit normal ,SGOT, SGPT, and ALP ≤ 3 x institutional upper limit normal
11. A patient who voluntarily signed a document for the study.

Exclusion Criteria:

1. Presumed FIGO stage III-IV
2. Neuroendocrine tumor histology
3. Other disease involving lymphatic system
4. lymphedema of the lower extremity or inguinal area
5. previous pelvic or paraaortic lymph node dissection
6. previous radiation or concurrent chemoradiation therapy of abdomen or pelvis
7. previous chemotherapy due to malignant disease of abdomen or pelvis
8. Patients who have had or have been treated for cancer within five years, other than non-melanoma skin cancer, carcinoma in situ of uterine cervix, stomach or bladder
9. severe, uncontrolled underlying diseases or underlying disease with complications
10. hypersensitivity to indocyanine green
11. a pregnant or breast-feeding woman

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 810 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
The 3-year disease-free survival (3-year DFS) | 3 years
  The time interval between the date of surgery and the date of recurrence will be caculated as month. The survival curve will be calculated suing Kaplan-Meir method, and survival difference will be compared using Log-rank test.

SECONDARY OUTCOMES:
Surgery-related morbidity rate | One month
  Compare the surgery-related morbidity rate after one month of surgery.
Incidence of lymphocele and lymphedema | 3 years
  After 3 years of surgery, the incidence of lymphocele and lymphedema are compared.
The 3-year overall survival (3-year OS) | 3 years
  The time interval between the date of surgery and the date of death of disease will be caculated as month. The survival curve will be calculated suing Kaplan-Meir method, and survival difference will be compared using Log-rank test.
The 5-year disease free survival (5-year DFS) | 5 years
  The time interval between the date of surgery and the date of recurrence will be caculated as month. The survival curve will be calculated suing Kaplan-Meir method, and survival difference will be compared using Log-rank test.
The 5-year overall survival (5-year OS) | 5-years
  The time interval between the date of surgery and the date of death of disease will be caculated as month. The survival curve will be calculated suing Kaplan-Meir method, and survival difference will be compared using Log-rank test.
The pattern of recurrence | 3 years
  Anatomic location of first recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lecuru F, Mathevet P, Querleu D, Leblanc E, Morice P, Darai E, Marret H, Magaud L, Gillaizeau F, Chatellier G, Dargent D. Bilateral negative sentinel nodes accurately predict absence of lymph node metastasis in early cervical cancer: results of the SENTICOL study. J Clin Oncol. 2011 May 1;29(13):1686-91. doi: 10.1200/JCO.2010.32.0432. Epub 2011 Mar 28. PMID 21444878
- [Background] Ballester M, Dubernard G, Lecuru F, Heitz D, Mathevet P, Marret H, Querleu D, Golfier F, Leblanc E, Rouzier R, Darai E. Detection rate and diagnostic accuracy of sentinel-node biopsy in early stage endometrial cancer: a prospective multicentre study (SENTI-ENDO). Lancet Oncol. 2011 May;12(5):469-76. doi: 10.1016/S1470-2045(11)70070-5. Epub 2011 Apr 12. PMID 21489874
- [Background] Bae HS, Lim MC, Lee JS, Lee Y, Nam BH, Seo SS, Kang S, Chung SH, Kim JY, Park SY. Postoperative Lower Extremity Edema in Patients with Primary Endometrial Cancer. Ann Surg Oncol. 2016 Jan;23(1):186-95. doi: 10.1245/s10434-015-4613-1. Epub 2015 May 19. PMID 25986870
- [Background] Tanner EJ, Sinno AK, Stone RL, Levinson KL, Long KC, Fader AN. Factors associated with successful bilateral sentinel lymph node mapping in endometrial cancer. Gynecol Oncol. 2015 Sep;138(3):542-7. doi: 10.1016/j.ygyno.2015.06.024. Epub 2015 Jun 19. PMID 26095896
- [Derived] Park JY, Kim JH, Baek MH, Park E, Kim SW. Randomized comparison between sentinel lymph node mapping using indocyanine green plus a fluorescent camera versus lymph node dissection in clinical stage I-II endometrial cancer: a Korean Gynecologic Oncology Group trial (KGOG2029/SELYE). J Gynecol Oncol. 2022 Nov;33(6):e73. doi: 10.3802/jgo.2022.33.e73. Epub 2022 Jul 25. PMID 36047376